CLINICAL TRIAL: NCT00605839
Title: Adapting Mobile Communication Technology to Improve the Management of Adolescents With Diabetes
Brief Title: Mobile Communication Technology for Adolescents With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Aaron Carroll, Assoc. Prof of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ADA-HenryBecton-DGM-01
Record Dates: First submitted 2008-01-17; First posted 2008-01-31 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes
Keywords: mobile technology; cell phones; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucopak Care (Experimental): Glucopak cell phone and intensive monitoring. This group will be given the experimental device, and placed in close communication with the clinic.
  Interventions: Device: GlucoPak
- Cell Phone Care (Active Comparator): Cell phone only, without the Glucopak. Participants will be given cell phones and encouraged to communicate more closely with the clinic, but will not use the Glucopak.
  Interventions: Device: Cell Phone
- Usual Care (Placebo Comparator): Usual care, without cell phone or glucopak
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: GlucoPak — We will be giving participants Glucopak devices and monitoring them closely over the 6 month period.
  Arms: Glucopak Care
Device: Cell Phone — We will provide cell phones and access to the clinic to facilitate communications
  Arms: Cell Phone Care
Other: Usual Care — This intervention was usual care, without either device.
  Arms: Usual Care

SUMMARY:
Among those with type I diabetes, adolescents can be among the worst at achieving glycemic control. Behaviors normal in adolescent development (e.g., developing independence, rejecting parental norms in favor of peers) can be at odds with the demands of effective diabetes self-management. Modifying the family and patient interaction should be a crucial component to improving the ability of an adolescent to manage his or her diabetes.

Mobile technology is becoming more popular in medicine, and adolescents, as a group are more inclined to accept technology as an adjunct to care. Mobile technology that links adolescents to health providers could help them to work through complex information that must be processed to make good decisions. Since this "assistance" comes from health professionals, it should help relax parents somewhat, thus reducing problems associated with parental hypervigilance and manipulation of the regimen to avoid problems of hypoglycemia. Parental-child conflicts may therefore be reduced by using cell phone glucose monitoring technology that directly reports self-blood glucose monitoring data to providers and creates a communication link to discuss therapeutic options.

This study investigates whether the use of mobile technology, in the form of a cell phone glucose monitoring system, will help reduce the need for parents to assert behavioral control, which can negatively impact adolescent diabetes self-management. The study will also determine whether adolescents report improved quality of life, demonstrate competence in diabetes management, and are able to achieve better control of their diabetes.

DETAILED DESCRIPTION:
Among patients with type I diabetes, adolescents struggle the most with self-management, which often results in poor glycemic control. Optimizing parent-patient interaction is crucial to improving self-management. Mobile technology with integrated glucose monitoring capability that links adolescents to providers may reduce parental hypervigilance and assist them to better understand self-management. .

This study will investigate a novel cell phone glucose monitoring system (CPGM) with the following specific aims:

1. To establish feasibility of a CPGM system as a component of an adolescent diabetes management program.
2. To determine if the technology will improve a) quality of parent-child relationship, b) patient quality of life, c) competence in diabetes management, and d) metabolic control.
3. To gather preliminary data for development of future intervention studies.

120 adolescents with type I diabetes will be randomly assigned to either an experimental or control group. Experimental subjects will use the CPGM which will transmit all blood glucose data to a host computer. A nurse practitioner in the pediatric endocrinology clinic will determine need for telephone contacts based on evaluation of transmitted data. Subjects might be telephoned to discuss possible regimen adjustments, need for clinic visits, or referrals to additional services. Subjects will also be able to initiate contact with the project nurse. Control subjects will continue to receive standard care. .

This study will assess the effect of the intervention in the four primary domains stated in the specific aims. These domains will be measured at baseline, three months, and six months.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent with thpe 1 diabetes
2. Adolescents in the study must intend to remain in the care of participating clinics for the extent of the study
3. Adolescents in the study must be literate in English.

Exclusion Criteria:

1. Only one patient per family can participate
2. Patients who participated in preliminary studies related to the development of the cell phone technology will be excluded.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Marrero, PhD, Principal Investigator — Indiana University School of Medicine; Aaron E Carroll, MD, MS, Study Director — Indiana University School of Medicine
Locations (1):
- Riley Hospital Diabetes Clinics, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the pediatric diabetes clinics at the James Whitcomb Riley Hospital for Children in Indianapolis, IN. Adolescents with type 1 diabetes between the ages of 14 and 18 years living with at least one parent participated.
Groups:
- Glucopak Cell Phone and Intensive Monitoring: Glucopak cell phone and intensive monitoring. Participants use the experimental device and are actively monitored by the clinic.
- Cell Phone Only: Cell phone only. Participants are given cell phones and encouraged to keep in contact with the clinic.
- Usual Care: Usual care, without Glucopak or cell phones.
Period: Overall Study
Arm/Group | Glucopak Cell Phone and Intensive Monitoring | Cell Phone Only | Usual Care
Started | 40 | 37 | 28
Completed | 39 (One patient would not keep to the text messaging constraints and had to be removed.) | 37 | 28
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Glucopak Cell Phone and Intensive Monitoring: Glucopak cell phone and intensive monitoring. This group will be given the experimental device, and placed in close communication with the clinic.
- Cell Phone Only: Cell phone only, without the Glucopak. Participants will be given cell phones and encouraged to communicate more closely with the clinic, but will not use the Glucopak.
- Total: Total of all reporting groups
Arm/Group | Glucopak Cell Phone and Intensive Monitoring | Cell Phone Only | Usual Care | Total
Number analyzed (Participants) | 40 | 37 | 28 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 37 | 28 | 105
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 13 | 53
  Male | 20 | 17 | 15 | 52
Region of Enrollment [Number; unit: participants]
  United States | 40 | 37 | 28 | 105

OUTCOME MEASURES:

1. Primary Outcome: Quality of Parent-child Relationship
Description: The Cornell Parent Behavior Description Scale was used to measure the antecedents and consequences of children's perceptions of the behavior of their parents towards them. Each of 14 subscales is scored from 0-10. The potential range of the total score is therefore 0 (fewest behaviors) to 140 (most behaviors). We used the total score, which is equivalent to the sums of the subscales, and calculated the change from baseline to 6 months. The range of the change is given as a 95% CI. A change of zero would indicate no change. A positive number is a worsening , and a negative number indicates an improvement.
Time Frame: Change from baseline to 6 months. Please see above for a description of how the change score should be interpreted.
Population: Everyone who completed the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Glucopak Cell Phone and Intensive Monitoring | Cell Phone Only | Usual Care
Number analyzed (Participants) | 39 | 37 | 28
units on a scale | 0.22 [-2.11 to 2.54] | -3.24 [-6.12 to -0.36] | -0.59 [-5.41 to 4.23]

ADVERSE EVENTS:
Arm/Group | Glucopak Cell Phone and Intensive Monitoring | Cell Phone Only | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 0/28
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 0/28

LIMITATIONS AND CAVEATS:
This was a small pilot study to generate results for further work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No